CLINICAL TRIAL: NCT07033052
Title: Developing Resilience and Anxiety Management Through the Arts (DRAMA) 2
Brief Title: Developing Resilience and Anxiety Management Through the Arts
Acronym: DRAMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Expanding Horizons Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20241298; NEA AWARD 1891861-38-22 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depression; Mood
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to participant condition in order to reduce assessor bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Improvisation + Wellness (Experimental): The Improvisation + Wellness arm will include a variety of techniques based on Cognitive Behavioral Therapy (CBT): behavior activation, mindfulness, relaxation techniques, exposure, and cognitive restructuring. The improvisation techniques will include using your truth (talk about what you know), making patterns (working with others in the group to create something that you all contribute to), yes…and (agreeing with others and building on what others contribute to activities/conversations).
  Interventions: Behavioral: Improvisation + Wellness
- Improvisation (Experimental): The improvisation alone arm involves the same improv techniques as the improv + wellness arm, but without the wellness techniques. Improv techniques include using your truth (talk about what you know), making patterns (working with others in the group to create something that you all contribute to), yes…and (agreeing with others and building on what others contribute to activities/conversations).
  Interventions: Behavioral: Improvisation
- Social Craft (Active Comparator): The social craft group involves youth connecting with other youth while completing craft projects.
  Interventions: Behavioral: Social Craft

INTERVENTIONS:
Behavioral: Improvisation + Wellness — Theatrical improvisation exercises, the theatrical art of performance and storytelling without a script, will be combined with wellness techniques
  Arms: Improvisation + Wellness
Behavioral: Improvisation — Theatrical improvisation exercises (the theatrical art of performance and storytelling without a script) will be completed in this arm. These exercises will be fairly similar to that from the improvisation + wellness but without the wellness techniques.
  Arms: Improvisation
Behavioral: Social Craft — Participants assigned to the Social Craft group will engage in arts and crafts projects and activities
  Arms: Social Craft

SUMMARY:
The Developing Resilience and Anxiety Management Through the Arts (DRAMA) Study examines the degree to which the arts can help to address stress, anxiety, and sad mood in children and adolescents. The researchers will pair theatrical improvisation exercises with cognitive-behavioral therapy (CBT) techniques versus improvisation exercises alone versus a social craft group on reducing elevated levels of anxiety and depression.

DETAILED DESCRIPTION:
The purpose of this study is to observe the benefits of theatrical improvisation exercises paired with cognitive-behavioral therapy (CBT) techniques versus improvisation exercises alone versus a craft control group on reducing elevated levels of anxiety and depression in children and adolescents. It is possible that improvisational techniques could reduce anxiety and depression symptoms because they involve being spontaneous and going into social situations as well as creating something larger than oneself through the group (e.g., creating a scene, working together, etc.). It is also possible that the addition of CBT techniques might lead to a further reduction in anxiety and depression. The study will compare these to a control craft group where youth work on craft projects. The researchers hypothesize that improvisation exercises paired with CBT techniques will be more effective at reducing anxiety and depression than improvisational exercises alone, which we expect will be more effective than a craft group. This improvisation course will not be implemented by licensed therapists or psychologists. Group leaders will be undergraduates, schoolteachers, and graduate students without a background in therapy or counseling (e.g., drama students, music students, etc.) As such, it is important to note that this should not be considered "therapy" or an "intervention." It should not replace intensive treatment for children or adolescents who require a higher level of treatment. Rather, it can be considered a supplementary or preventative group that can help children or adolescents manage feelings of anxiety or depression. The goal of the study is to reduce existing levels of anxiety and depression, prevent the development of new symptoms, and prevent exacerbation of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 17 years of age
* Individuals must have parental/guardian consent
* Elevated levels of anxiety or depression based on

  1. Screen for Child Anxiety Related Disorders (SCARED) score of 15 or higher, or;
  2. Revised Children's Anxiety and Depression Scale (RCADS) Depression T score of 65 or higher, or;
  3. Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) clinician severity rating of 3 on any anxiety disorder or on a mood-related disorder

Exclusion Criteria:

* Diagnosed with Conduct Disorder or with behavioral symptoms that would make it difficult for the child/adolescent to participate in the group or comply with directions given by the group leader (such as difficulty following instructions, difficulty staying in one's seat, defiance of adults, harming animals or people, threatening others, getting into physical fights, hyperactivity, impulsivity, difficulty waiting for one's turn, etc.)
* Autism or developmental delays
* Psychotic symptoms or active suicidality
* Active Eating Disorders that raise concerns about morbidity and therefore need to be addressed in an intervention and actively monitored
* Unsteady dosage or recently or impending changes to psychotropic medication(s)
* Non-English-speaking individuals
* Wards of the State

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Child Anxiety and Depression (based on Parent Report) | Baseline, post (after 9 weeks of the group curriculum), and 3 months post-group
  Child anxiety and depression will be measured using a parent-report. The Revised Child Anxiety and Depression Scale Parent Report (RCADS-P) is a 47-item measure that assesses parent-report of child anxiety and depressive symptoms. Parents respond to each item on a 4-point Likert-scale from 0 ("never") to 3 ("always). The measure yields 6 subscales including: separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). There is also a total anxiety scale, which is the sum of the 5 anxiety subscales and a total internalizing scale, which is the sum of all 6 subscales. The RCADS-P has excellent psychometric properties, including high internal consistency and convergent validity. Higher scores indicate higher anxiety/depression symptoms. A T-score is created based on the child's age and gender.
Child Anxiety and Depression (based on youth report) | Baseline, post (after 9 weeks of the group curriculum), and 3 months post-group
  Child anxiety and depression will also be measured using a youth report. The Revised Child Anxiety and Depression Scale (RCADS) is a 47 item measure that assesses child report of child anxiety and depressive symptoms. Youth respond to each item on a 4-point Likert-scale from 0 ("never") to 3 ("always). The measure yields 6 subscales including: separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). There is also a total anxiety scale, which is the sum of the 5 anxiety subscales and a total internalizing scale, which is the sum of all 6 subscales. The RCADS has been translated from English into Spanish, Chinese, Dutch, and Danish. The measure has good discriminant validity, internal consistency, and convergent validity and discriminates between anxiety and depression.
Cognitive Behavioral Technique (CBT) Skill Knowledge | Baseline, after 9 weeks of the group curriculum, and 3 months post-group
  This is a measure designed by the research team that assesses cognitive-behavioral techniques (CBT) Skills knowledge. Participants indicate whether each item is true or false. Items ask about whether thoughts and feelings influence one another, whether avoidance is a good idea when one is anxious about something, present-moment focus/mindfulness, diaphragmatic breathing, activity scheduling, progressive muscle relaxation, etc.
Cognitive Behavioral Technique (CBT) Skills Use | Baseline, after 9 weeks of the group curriculum, and 3 months post-group
  This is a measure designed by the research team that assesses cognitive-behavioral technique (CBT) Skills use. Participants indicate how often they use each skill on a scale from Never (0) to At least once a day (5). Skills assessed included diaphragmatic breathing, cognitive restructuring, facing your fears, muscle relaxation, being mindful, scheduling pleasant activities, etc.

SECONDARY OUTCOMES:
Youth mindfulness | Baseline, post (after 9 weeks of the group curriculum), and 3 months post-group
  Youth mindfulness will be measured using the Child and Adolescent Mindfulness Measure. The Child and Adolescent Mindfulness Measure (CAMM) is a youth report measure that assesses present-moment awareness and non-judgmental responses to internal experiences. Youth rate each item on a five-point Likert scale ranging from 0 ("never true") to 4 "always true." The scale yields a total score with lower scores indicating greater mindfulness. Internal consistency of the scale is strong (α = .81-.84) and it correlates negatively with internalizing, externalizing, somatic symptoms.
Connectedness | Baseline, post (after 9 weeks of the group curriculum), and 3 months post-group
  Youth will complete the Hemingway Measure of Adolescent Connectedness, which is a measure of connectedness across multiple spheres (neighborhood, friends, self-in-the-present, parents, siblings, school, peers, teachers, future, reading, kids from other cultures, religion, romantic partner, mother, and father). This study will only include the friends, self-in-the-present, parents, peers, and future subscales. Participants rate each item on how accurate it is on a Likert scale ranging from Not true (1), Sort of True(2), True (3), and Very True (4). Higher scores indicate greater connectedness within the particular sphere that the subscale is measuring.
Emotion regulation | Baseline, post (after 9 weeks of the group curriculum), and 3 months post-group
  Difficulties in Emotion RegulationScale (DERS) is a 36-item measure of emotion regulation in adults and youth. Participants rate how frequently they experience each item on a scale of 1 (almost never), 2 (sometimes), 3 (about half the time), 4 (most of the time), 5 (almost always). The DERS consists of the 6 subscales: emotional clarity, emotional awareness, goal-orientation in the presence of distress, perceived access to ER strategies, ability to control impulsive behavior in the presence of distress, and nonacceptance of emotions. Higher scores indicate higher levels of difficulties in the particular type of emotion regulation difficulty assessed by each subscale.
  The measure has been used in children and adolescents across a variety of ages and has good psychometric properties including good internal consistency, test-retest reliability, adequate construct, and predictive validity.
Self-esteem | Baseline, after 9 weeks of the group curriculum, and 3 months post-group
  Self-Esteem will be measured by The Rosenberg Self-Esteem Scale (RSES), a tool consisting of 10 statements rated on a four-point Likert scale. Each statement is rated on a scale from 0 to 3, with higher scores indicating higher self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Przeworski, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States